CLINICAL TRIAL: NCT05705362
Title: Randomized Controlled Trial of Simple CROSSsover Versus Side Branch Opening on Clinical Outcomes in Patients With Non-Left Main BIfurcation LeSion (CROSS-COBIS)
Brief Title: Simple Crossover Versus Side Branch Opening in Patients With Non-Left Main Bifurcation Lesion
Acronym: CROSS-COBIS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Keimyung University Dongsan Medical Center (Other)
Responsible Party: Principal Investigator, NAM, Chang-Wook, Professor, Keimyung University Dongsan Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CROSS-COBIS
Record Dates: First submitted 2022-12-19; First posted 2023-01-30 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Coronary Artery Disease
Keywords: Percutaneous coronary intervention; Bifurcation; Treatment strategy; Side branch
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Simple crossover arm (Experimental): This arm will receive the main vessel stenting only (with proximal optimization technique).
  Interventions: Procedure: Simple Crossover
- Side branch opening arm (Active Comparator): This arm will receive a side branch opening procedure after the main vessel stenting.
  Interventions: Procedure: Side branch opening

INTERVENTIONS:
Procedure: Simple Crossover — Regardless of allocated arms, stent implantation in the MV (selected 1:1 according to the distal MV size) followed by systematic proximal optimization technique (POT, post-dilatation of the stent at the level of proximal MV with a balloon diameter sized 1:1 according to the proximal MV) or POT like procedure is strongly recommended.
  Arms: Simple crossover arm
Procedure: Side branch opening — According to the latest European Bifurcation Club (EBC) consensus document, distal SB rewiring followed by kissing balloon inflation (eventually conducted with short non-compliant balloons) and repeat POT procedures are highly recommended. An additional stent will be allowed if major dissection or decreased TIMI flow of SB occurs during SB treatment.
  Arms: Side branch opening arm

SUMMARY:
Hypothesis:

Simple crossover strategy would be non-inferior to SB opening strategy in the risk of target lesion failure (TLF) in patients with angiographically compromised SB (visually SB stenosis ≥50%) after provisional MV stenting for non-left main bifurcation lesion.

A total of 1000 patients (500 per each group) with the angiographically compromised SB (visually SB stenosis ≥50%) after provisional MV stenting for non-left main bifurcation lesion will be enrolled. Patients will be randomized to either the simple crossover strategy group or SB opening strategy group at the time of enrollment with 1:1 ratio. Stratified randomization according to participating center, clinical presentation (acute coronary syndrome or stable ischemic heart disease), and type of bifurcation lesions (true or non-true) will be performed.

DETAILED DESCRIPTION:
Despite advances in stenting techniques and devices, percutaneous coronary intervention (PCI) for bifurcation lesions remains one of the most challenging and complex procedures. Current guidelines recommend 1-stenting with provisional side branch (SB) approach should be an initial treatment strategy for the bifurcation lesions, based on the previous results of several randomized trials. However, the standardization of the provisional strategy is limited. In particular, there is a recommendation on the treatment technique for SB when SB intervention is required, but It has not been decided in which cases SB treatment is necessary, in the latest European Bifurcation Club (EBC) consensus document.16 In previous studies, the criteria for performing SB opening after MV stent intervention in the 1-stenting with provisional SB approach were varied. In the DK-CUSH II (Double Kissing Crush versus Provisional Stenting Technique for Treatment of Coronary Bifurcation Lesions) or CACTUS (Coronary Bifurcations: Application of the Crushing Technique Using Sirolimus-Eluting Stents) trials, SB intervention was performed when the SB diameter stenosis more than 50%, grade B or higher dissection, or blood flow disturbance (TIMI flow 2 or less) after MV stent insertion. On the other hand, in the Nordic trial, the authors applied strict criteria for SB intervention after MV stent insertion (TIMI flow 2 or less only). Furthermore, there have been conflicting results regarding the clinical and angiographic outcomes of the jailed SB opening strategy after the main vessel (MV) stenting, compared with the simple crossover strategy for non-left main bifurcation lesion.

On this background, this trial aims to compare the clinical outcomes between simple crossover and side branch opening strategies in patients with the angiographically compromised SB (visually SB stenosis ≥50%) after provisional MV stenting for non-left main bifurcation lesion.

ELIGIBILITY:
Inclusion Criteria:

* (1) Subject must be at least 19 years of age
* (2) Patients with non-left main bifurcation lesion (SB diameter ≥2.3 mm)
* (3) Target lesions amenable for 1-stenting with provisional SB approach by operators' decision
* (4) Angiographically compromised SB (visual SB stenosis ≥50%) after provisional MV stenting

Exclusion Criteria:

* (1) Target lesions requiring elective 2-stenting technique by operators' decision (Observation Group 1)*
* (2) Patients who inevitably require SB intervention after MV stenting, as follows. (Observation Group 2)*

  1. Reduced SB TIMI flow (≤2) after MV stenting
  2. SB dissection after MV stenting (≥ Type C)
* (3) Patients without SB compromise after MV stenting (visually SB stenosis <50%) (Observation Group 3)*
* (4) Cardiogenic shock (Killip class IV) at presentation
* (5) Patients with significant valvular heart disease or severe left ventricular systolic dysfunction (ejection fraction <35%)
* (6) Pregnancy or breast feeding
* (7) Non-cardiac co-morbid conditions are present with life expectancy <1 year or that may result in protocol non-compliance (per site investigator's medical judgment)
* (8) Unwillingness or inability to comply with the procedures described in this protocol

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2023-03-01 (Estimated); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Target-lesion failure | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  a composite of cardiac death, myocardial infarction, and target-lesion revascularization

SECONDARY OUTCOMES:
All-cause death | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Death from any causes
Cardiac death | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Death from cardiac causes
Myocardial infarction | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  any myocardial infarction
Target-vessel myocardial infarction | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  myocardial infarction in target-vessel
Target-lesion revascularization | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Clinically indicated target-lesion revascularization
Target-vessel revascularization | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Clinically indicated target-vessel revascularization
Any revascularization | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Repeat revascularization procedure
Stent thrombosis | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  definite or probable stent thrombosis by Academic Research Consortium [ARC] definition
Bleeding | up to 2 years of median follow-up (till 1 year after the last patient enrollment)
  Bleeding ARC type 2, 3 or 5 bleeding
Total procedure time | at 1 day
  procedure time
Total amount of contrast use | at 1 day
  used contrast amount
Incidence of contrast induced nephropathy | 72 hours after the index procedure
  defined as an increase in creatinine of ≥0.5mg/dL or ≥25% from baseline within 72 hours after contrast exposure

IPD SHARING:
Plan to Share IPD: Undecided